CLINICAL TRIAL: NCT06902324
Title: Wild Mushroom Poisoning: a Case Series from Himalaya District
Status: Completed | Type: Observational
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Sishir Poudel, Principal Investigator, B.P. Koirala Institute of Health Sciences
Other Study IDs: Ref No. 397
Record Dates: First submitted 2025-03-10; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Poisoning Patients

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Introduction: Mushroom poisoning is a significant yet underreported issue in Nepal, particularly in rural areas where wild mushrooms are a vital food source. Poisonous mushrooms, often indistinguishable from edible species, pose severe health risks.

Case reports: This case series documents ten patients (6 males, 4 females) aged 19 to 39 from Mustang, Nepal, who developed symptoms of cholinergic toxicity approximately one hour after consuming wild mushrooms collected from a high-altitude region. Common symptoms included blurry vision (80%), vomiting (60%), sweating (50%), and abdominal pain (20%). A notable case involved a 19-year-old female who exhibited severe symptoms, including hypotension, tachycardia, and respiratory distress, requiring atropine therapy. All patients were managed with supportive care, including intravenous fluids and symptomatic treatments, and recovered fully within 12 hours.

Keywords: Cholinergic; Muscarinic; Toxidrome; Toxin

DETAILED DESCRIPTION:
Introduction Mushroom poisoning can present with a wide range of clinical features, including gastrointestinal distress, neurotoxicity, myotoxicity, metabolic disturbances, and severe outcomes such as liver and kidney failure.These poisonings are most frequent during the spring and autumn seasons, as the cool, damp evenings in these periods promote mushroom growth. Non-toxic and toxic mushrooms often grow in close proximity, and many poisonous species are difficult to distinguish from edible ones, increasing the risk of accidental ingestion.

The growing popularity of mushroom consumption has contributed to a rise in poisoning cases. This is often attributed to difficulties in distinguishing toxic species, accidental ingestion of nearby poisonous mushrooms, improper cooking methods, or contamination with bacteria or viruses.

Nepal is home to a diverse range of mushrooms, with 159 edible species, 74 medicinal species, and 100 known poisonous species. Mushroom poisoning is a recurring issue in the country, leading to dozens of deaths and hundreds of hospitalizations annually, with many others relying on local treatments.

During the rainy season, the dependency on wild mushrooms increases among poorer communities, who often use them as a vital food source. Although locals possess significant knowledge of wild mushrooms, tragic accidents still occur, sometimes resulting in the loss of entire families. Many individuals remain confident in their ability to identify toxic mushrooms despite having witnessed fatalities. The lack of documentation for numerous poisoning incidents in remote areas highlights the need to preserve and record traditional knowledge before it is lost.

This case series provides essential data to address gaps in literature regarding toxicological effects of specific mushroom, supporting clinicians and researchers. It also encourages further studies in clinical medicine, toxicology, mycology, and public health to improve management and awareness of mushroom-related risks.

ELIGIBILITY:
Inclusion Criteria:

* Consumed wild mushroom

Exclusion Criteria:

* Didn not consume wild mushroom

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants consuming wild mushroom
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Death | Baseline
  Yes/No

CONTACTS AND LOCATIONS:
Locations (1):
- Mustang Hospital, Jomsom, Nepal

IPD SHARING:
Plan to Share IPD: No